CLINICAL TRIAL: NCT03242915
Title: Phase II Study of Pembrolizumab in Combination With Platinum-based Chemotherapy in Nonsmall Cell Lung Cancer Patients With Targetable Genetic Alterations Previously Treated With Appropriate Targeted Agents With Progressive Disease
Brief Title: Pembrolizumab Plus Chemotherapy in NSCLC With Targetable Genetic Alterations After Progression on Targeted Agents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2017.057; HUM00129169 (Other: University of Michigan)
Record Dates: First submitted 2017-08-03; First posted 2017-08-08 (Actual); Results first posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab/Carboplatin/Pemetrexed (Experimental): Pembrolizumab 200 mg with carboplatin at AUC (area under the curve dosing) 5 and pemetrexed at 500 mg/m2 administered intravenously every 3 weeks
  Interventions: Drug: Pembrolizumab; Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: Pembrolizumab — 200mg IV every 3 weeks
Drug: Carboplatin — AUC 5 IV every 3 weeks
Drug: Pemetrexed — 500 mg/m^2 IV every 3 weeks

SUMMARY:
Investigators hypothesize that addition of pembrolizumab will enhance the efficacy of carboplatin and pemetrexed in patients with EGFR-mutation-positive NSCLC, or patients with other genetic alterations, and who have disease progression following appropriate targeted therapies.

ELIGIBILITY:
Inclusion Criteria:

* Cohort-specific:

Cohort 1- EGFR mutation positive NSCLC patients previously treated with appropriate targeted therapy with progressive and measurable disease per RECIST 1.1 criteria tumor.

Cohort 2- Other genetically altered NSCLC patients previously treated with appropriate targeted therapy with progressive and measurable tumor.

* Tumor tissue for PD-L1 assessment should be available unless PD-L1 assessment results are already available.
* Patients should not have received any systemic chemotherapy for advanced NSCLC. Patients who received 1 cycle of systemic chemotherapy for advanced NSCLC while awaiting the results of tumor molecular analysis and subsequently were switched to appropriate targeted therapy will be eligible. Patients who have received neoadjuvant, adjuvant or as part of concurrent chemotherapy and radiation are eligible if they received the chemotherapy 12 months or more before the start of study therapy.
* ECOG PS 0-1 (Eastern Cooperative Oncology Group Performance Status: an attempt to quantify cancer patients' general well-being and activities of daily life. The score ranges from 0 to 5 where 0 is asymptomatic and 5 is death.)
* Patients should have recovered to ≤ grade 1 from clinically meaningful (example alopecia is not considered clinically meaningful) adverse events related to prior treatments.
* Patients should be willing and able to provide written informed consent for the trial.
* Be ≥ 18 years of age on day of signing informed consent.
* Demonstrate adequate organ function
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 1 week of enrollment.
* Female subjects of childbearing potential must be willing to use an adequate method of contraception
* Male subjects of child bearing potential must agree to use an adequate method of contraception

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment. If the half-life of the drug is known then starting therapy 5 half-lives after the end of the last therapy is acceptable.
* Has a diagnosis of immunodeficiency. Patient should not be of any immunosuppressive therapy or steroids > prednisone 10mg/day or its equivalent on the day of the start of therapy.
* Has a known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab, carboplatin or pemetrexed or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had targeted small molecule therapy, or palliative radiation therapy within 1 week prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
* Has a known additional malignancy that is progressing or requires active treatment or the treating physician believes will require therapy within 1 year.
* Has symptomatic central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has active autoimmune disease that has required systemic treatment in the past 2 years
* Has known history of non-infectious pneumonitis that required steroids or has current pneumonitis. Has known history of interstitial lung disease.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B or Hepatitis C
* Has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Kalemkerian, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (7):
- United States (7):
  - Rush University Medical Center, Chicago, Illinois
  - The University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Cancer Institute/Henry Ford Hospital, Detroit, Michigan
  - Montefiore Cancer Center, The Bronx, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Sarah Cannon, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- EGFR+ NSCLC; ALK+ NSCLC: Pembrolizumab 200 mg with carboplatin at AUC (area under the curve dosing) 5 and pemetrexed at 500 mg/m2 administered intravenously every 3 weeks
  Pembrolizumab: 200mg IV every 3 weeks
  Carboplatin: AUC 5 IV every 3 weeks
  Pemetrexed: 500 mg/m^2 IV every 3 weeks
Period: Overall Study
Arm/Group | EGFR+ NSCLC | ALK+ NSCLC
Started | 26 | 7
Completed | 17 | 3
Not Completed | 9 | 4
Not completed — Adverse Event | 5 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Physician Decision | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EGFR+ NSCLC | ALK+ NSCLC | Total
Number analyzed (Participants) | 26 | 7 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 3 | 14
  >=65 years | 15 | 4 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 4 | 21
  Male | 9 | 3 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 21 | 6 | 27
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 0 | 4
  White | 17 | 6 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 26 | 7 | 33

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients That Respond to Treatment
Description: The primary endpoint is Response Rate (RR) defined as the rate of complete and partial response. Complete Response (CR): Disappearance of all non-target lesions. All lymph nodes must be non-pathological in size (<10mm short axis). Partial Response (PR): Persistence of one or more non-target lesion(s) but does not qualify for PD. Progressive Disease (PD): Unequivocal progression of existing non-target lesions. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: 5.5 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | EGFR+ NSCLC | ALK+ NSCLC
Number analyzed (Participants) | 26 | 7
percentage of patients | 46 [27 to 67] | 29 [4 to 71]

2. Secondary Outcome: Progression Free Survival (PFS) Time
Description: PFS is defined as the duration of time from registration to time of progression. Progressive Disease (PD): Unequivocal progression of existing non-target lesions. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: 5.5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | EGFR+ NSCLC | ALK+ NSCLC
Number analyzed (Participants) | 26 | 7
Months | 8.3 [7.2 to 16.5] | 2.9 [1.1 to NA] — Not evaluable as there were not a sufficient number of events for us to estimate those values

3. Secondary Outcome: Overall Survival (OS) Time
Description: Overall survival is defined as the time from registration to time of death. If the patient is lost to follow-up, survival will be censored on the last date the patient was known to be alive.
Time Frame: 5.5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | EGFR+ NSCLC | ALK+ NSCLC
Number analyzed (Participants) | 26 | 7
Months | 22.2 [20.6 to NA] — Not evaluable as there were not a sufficient number of events for us to estimate those values | 2.9 [1.1 to NA] — Not evaluable as there were not a sufficient number of events for us to estimate those values

ADVERSE EVENTS:
Time Frame: All adverse event data (serious and non-serious) collected from the time of the initial study treatment administration through 30 days (non-serious) and 90 days (serious) after the last dose of study treatment. Up to 2 years for adverse events and serious adverse events. 5.5 years for survival.
Arm/Group | EGFR+ NSCLC | ALK+ NSCLC
All-Cause Mortality (participants affected / at risk) | 24/26 | 7/7
Serious Adverse Events (participants affected / at risk) | 10/26 | 7/7
Other Adverse Events (participants affected / at risk) | 26/26 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EGFR+ NSCLC (N=26) | ALK+ NSCLC (N=7)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Acidosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Back pain (General disorders) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Investigations) | 0 (0) | 1 (1)
Progressive Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1) — C. diff
Lung infection (Infections and infestations) | 2 (2) | 1 (1)
Pericardial tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Pleural effusion (Infections and infestations) | 0 (0) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Stroke (General disorders) | 1 (1) | 0 (0)
Thromboembolic event (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EGFR+ NSCLC (N=26) | ALK+ NSCLC (N=7)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 11 (22) | 1 (1)
Alkaline phosphatase increased (Investigations) | 7 (10) | 2 (2)
Allergic reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alopecia (General disorders) | 1 (1) | 0 (0)
Amnesia (General disorders) | 1 (1) | 0 (0)
Anemia (Investigations) | 21 (46) | 5 (18)
Anorexia (Metabolism and nutrition disorders) | 7 (9) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1)
Arthralgia (General disorders) | 3 (3) | 0 (0)
Arthritis (General disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 8 (14) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Back pain (General disorders) | 3 (3) | 0 (0)
Blood bilirubin increased (Renal and urinary disorders) | 2 (3) | 1 (1)
Blurred vision (Eye disorders) | 3 (3) | 0 (0)
Bone pain (General disorders) | 4 (4) | 1 (1)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0)
Cholesterol high (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2) | 1 (1)
Conjunctivitis (Eye disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 13 (18) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 1 (1)
Creatinine increased (Investigations) | 5 (8) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 4 (5) | 1 (1)
Depression (Psychiatric disorders) | 3 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 5 (6) | 3 (3)
Dizziness (General disorders) | 5 (9) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Dysgeusia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (General disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 1 (1)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Tenderness
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1) | 0 (0) — fullness
Edema face (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 6 (7) | 2 (2)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (1) | 0 (0) — cold intolerance
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (1) | 0 (0) — Diabetes Insipidus
Epistaxis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Double Vision
Facial pain (General disorders) | 1 (1) | 0 (0)
Fall (General disorders) | 2 (7) | 0 (0)
Fatigue (General disorders) | 17 (24) | 5 (10)
Fever (General disorders) | 4 (4) | 1 (1)
Flu like symptoms (General disorders) | 1 (1) | 0 (0)
Flushing (General disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 0 (0) — polydipsia
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 1 (1) — Night sweat
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (3) | 2 (2)
Headache (Nervous system disorders) | 4 (5) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (22) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 5 (5) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (9) | 4 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (8) | 2 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 6 (10) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 14 (18) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 3 (4) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Infusion related reaction (General disorders) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (1) | 0 (0) — Grey stool
Investigations - Other, specify (Investigations) | 0 (0) | 1 (1) — Low protien
Investigations - Other, specify (Investigations) | 0 (0) | 1 (1) — TSH increased
Investigations - Other, specify (Investigations) | 0 (0) | 1 (1) — Leucocytosis
Irritability (General disorders) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 10 (36) | 5 (11)
Malaise (General disorders) | 1 (1) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (2) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 15 (20) | 5 (7)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Left eye Cyst
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Excision of left axillary cyst
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 0 (0) — Syncope
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 0 (0) — Brain fog
Neutrophil count decreased (Investigations) | 9 (21) | 1 (1)
Non-cardiac chest pain (General disorders) | 3 (3) | 2 (2)
Pain (General disorders) | 8 (11) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 6 (10) | 2 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — tachypnea
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Dysphonia
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus pain (Nervous system disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 4 (5) | 4 (6)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Rash NOS
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 3 (4)
Upper respiratory infection (Infections and infestations) | 3 (4) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (7) | 4 (5)
Watering eyes (Eye disorders) | 3 (5) | 0 (0)
Weight gain (Investigations) | 1 (2) | 0 (0)
Weight loss (Investigations) | 5 (5) | 2 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
White blood cell decreased (Investigations) | 15 (44) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
* Participating Sites agree not to publish or publicly present the Study Data or Study Results until Michigan or Michigan's Principal Investigator have first Published the Study Data or Study Results
* All Study Data and Results generated by the Participating Site will be owned by Participating Site
* Sponsors have the right to review and comment on any Public Presentation as defined by the contract
* Other limitations outline within the contract

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-03): https://cdn.clinicaltrials.gov/large-docs/15/NCT03242915/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/15/NCT03242915/ICF_001.pdf